CLINICAL TRIAL: NCT01243957
Title: LY2216684 and Fluoxetine Pharmacokinetic Interaction Study in Healthy Subjects
Brief Title: A Study to Measure if There is Any Difference in How the Body Breaks Down or Inactivates Either Fluoxetine or LY2216684 When Both of These Medicines Are Given Together.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12597; H9P-EW-LNCH (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2216684 + fluoxetine (Experimental): LY2216684: 18 milligrams (mg) oral (po) once daily (QD) on Days 1, 2, and 3 and Days 25-27
  Fluoxetine: 60 mg po QD for 7 days (Days 4-10) then 20 mg po QD for 17 days (Days 11-27)
  Interventions: Drug: LY2216684; Drug: Fluoxetine

INTERVENTIONS:
Drug: LY2216684 — LY2216684: 18 mg po QD on Days 1, 2, and 3 and Days 25-27
Drug: Fluoxetine — Fluoxetine: 60 mg po QD for 7 days (Days 4-10) then 20 mg po QD for 17 days (Days 11-27)

SUMMARY:
The purpose of this study is to measure if there is any difference in how the body breaks down or inactivates either fluoxetine or LY2216684 when both of these medicines are given together. This study will look at how fluoxetine might affect LY2216684 and how giving LY2216684 might affect fluoxetine in the body.

The duration of study participation in this study is approximately 36 days not including the screening appointment. This study requires 1 research unit confinement of 29 days/28 nights followed by 1 outpatient appointment. A screening appointment is required within 30 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical history and physical examination.
* Male participants: Agree to use a reliable method of birth control during the study + 3 months following the last dose of study drug.
* Female participants: Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control for 6 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study + 1 month following the last dose of study drug; or are women not of child-bearing potential due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation) or menopause (at least 1 year without menses or 6 months without menses and a follicle stimulating hormone (FSH) level ≥40 mass International Units per milliliter (mIU/mL).
* Are between the ages of 18-65 years, inclusive.
* Are between the body mass index (BMI) of 18.5-32.0 kilograms per square meter (kg/m^2), inclusive.
* Have screening clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have venous access sufficient to allow blood sampling according to the protocol.
* Have normal blood pressure (BP) and pulse rate (supine position and standing) as determined by the investigator.
* Are reliable and available for the duration of the study and are willing to follow study procedures.
* Provided written informed consent approved by Lilly and the institutional review board (IRB) governing the site.

Exclusion Criteria:

* Are investigator site personnel directly affiliated with this study or their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
* Are Lilly employees.
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device other than the study drug used in this study, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to LY2216684, fluoxetine, or related compounds.
* Are persons who previously completed or discontinued from this study, or any other study investigating LY2216684 within 6 months prior to screening.
* Have a clinically significant abnormality in the 12-lead electrocardiogram (ECG) as determined by the investigator.
* Have significant history of or current cardiovascular (including dysrhythmias), respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have a history of seizure disorders.
* Have a history or presence of the signs and/or symptoms of hyponatremia.
* Have a history or presence of the signs and/or symptoms of hyperthyroidism as determined by an abnormal thyroid stimulating hormone (TSH) at screening.
* Show evidence of significant active neuropsychiatric disease or a history of suicidal thoughts or attempted suicide.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Are women with a positive pregnancy test or women who are lactating.
* Intend to use over-the-counter or prescription medication within 14 days prior to dosing, unless deemed acceptable by the investigator and sponsor's medical monitor.
* Use of any drugs or substances that are known to be a strong inducer or inhibitor of cytochrome P450 2D6 (CYP2D6) within 30 days prior to check-in.
* Have donated blood of more than 500 milliliters (mL) within 4 weeks prior to screening.
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption 48 hours prior to check-in until the completion of the study (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any participants unwilling to adhere to study caffeine restrictions.
* Have used any tobacco-containing or nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to enrollment.
* Have consumed grapefruit or grapefruit-containing products 7 days prior to enrollment and during the study.
* Have a documented or suspected history of glaucoma.
* Participants are determined to be unsuitable by the investigator for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Evansville, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2216684 + Fluoxetine: LY2216684: 18 milligrams (mg) oral (po) once daily (QD) on Days 1-3 and Days 25-27.
  Fluoxetine: 60 mg po QD for 7 days (Days 4-10) then 20 mg po QD for 17 days (Days 11-27).
Period: Overall Study
Arm/Group | LY2216684 + Fluoxetine
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LY2216684 + Fluoxetine
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Plasma Concentration-Time Curve Over a 24-Hour Dosing Interval (AUCτ) of LY2216684
Description: The Least Squares (LS) geometric mean AUCτ of LY2216684 was calculated based on the LY2216684 plasma concentration time curve from time 0 hour (hr) to time 24 hr (tau [τ]) when LY2216684 was administered alone (Day 3) and when LY2216684 was coadministered with fluoxetine (Day 27). The Day 27-to-Day 3 ratio of the LY2216684 LS geometric mean of AUCτ and the associated 90% confidence interval (CI) of the ratio were calculated.
Time Frame: Predose and 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Days 3 and 27
Population: The safety population included participants who were randomized, received study drug, and had at least 1 postdose safety assessment.
Measure: Least Squares Mean (90% Confidence Interval); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | LY2216684 + Fluoxetine
Number analyzed (Participants) | 20
hour*nanogram per milliliter (h*ng/mL)
  LY2216684 alone | 677 [609 to 753]
  LY2216684 + fluoxetine | 1210 [1090 to 1350]
Statistical Analysis 1: Comparison: LY2216684 + Fluoxetine; Test type: Superiority or Other; ANOVA; Ratio of Geometric LS Means = 1.79, 90% CI 2-sided [1.61 to 2.00]

2. Primary Outcome: Pharmacokinetic (PK) Parameter: Maximum Plasma Concentration (Cmax) of LY2216684
Description: The Least Squares (LS) geometric mean Cmax of LY2216684 was determined when LY2216684 was administered alone (Day 3) and when LY2216684 was coadministered with fluoxetine (Day 27). The Day 27-to-Day 3 ratio of the LY2216684 LS geometric mean of Cmax and the associated 90% confidence interval (CI) of the ratio were calculated.
Time Frame: Predose and 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Days 3 and 27
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Arm/Group | LY2216684 + Fluoxetine
Number analyzed (Participants) | 20
nanogram per milliliter (ng/mL)
  LY2216684 alone | 55.5 [50.8 to 60.7]
  LY2216684 + fluoxetine | 90.6 [82.8 to 99.0]
Statistical Analysis 1: Comparison: LY2216684 + Fluoxetine; Test type: Superiority or Other; ANOVA; Ratio of Geometric LS Means = 1.63, 90% CI 2-sided [1.49 to 1.79]

3. Primary Outcome: Pharmacokinetic (PK) Parameter: Time to Maximum Plasma Concentration (Tmax) of LY2216684
Description: Tmax of LY2216684 was determined using the median of paired differences between the 2 treatment groups when LY2216684 was administered alone (Day 3) and when LY2216684 was coadministered with fluoxetine (Day 27). The 90% confidence interval (CI) for the median of differences was calculated.
Time Frame: Predose and 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Days 3 and 27
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | LY2216684 + Fluoxetine
Number analyzed (Participants) | 20
hours
  LY2216684 alone | 3.00 [1.00 to 6.00]
  LY2216684 + fluoxetine | 3.00 [2.00 to 4.07]
Statistical Analysis 1: Comparison: LY2216684 + Fluoxetine; Test type: Superiority or Other; p = 0.5459, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-0.50 to 0.50]

4. Secondary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Plasma Concentration Time-Curve Over a 24-Hour Dosing Interval (AUCτ) of Fluoxetine and Norfluoxetine
Description: The Least Squares (LS) geometric means AUCτ of fluoxetine and norfluoxetine were calculated based on the fluoxetine and norfluoxetine plasma concentration time curves from time 0 hour (hr) to time 24 hr (tau [τ]) when fluoxetine was administered alone (Day 24) and when fluoxetine was coadministered with LY22166684 (Day 27). The Day 27-to-Day 24 ratios of fluoxetine and norfluoxetine LS geometric means of AUCτ and the associated 90% confidence interval (CI) of the ratios were calculated.
Time Frame: Predose and 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Days 24 and 27
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | LY2216684 + Fluoxetine
Number analyzed (Participants) | 20
hour*nanogram per milliliter (h*ng/mL)
  fluoxetine alone | 3450 [3060 to 3890]
  fluoxetine + LY2216684 | 3500 [3100 to 3940]
  norfluoxetine alone | 3170 [2790 to 3590]
  norfluoxetine + LY2216684 | 3280 [2890 to 3720]
Statistical Analysis 1: Comparison: LY2216684 + Fluoxetine; Ratio of Geometric LS Means of AUCτ for fluoxetine alone and fluoxetine + LY2216684; Test type: Superiority or Other; ANOVA; Ratio of Geometric LS Means = 1.01, 90% CI 2-sided [0.99 to 1.04]
Statistical Analysis 2: Comparison: LY2216684 + Fluoxetine; Ratio of Geometric LS Means of AUCτ for norfluoxetine alone and norfluoxetine + LY2216684; Test type: Superiority or Other; ANOVA; Ratio of Geometric LS Means = 1.04, 90% CI 2-sided [1.01 to 1.06]

5. Secondary Outcome: Pharmacokinetic (PK) Parameter: Maximum Plasma Concentration (Cmax) of Fluoxetine and Norfluoxetine
Description: The Least Squares (LS) geometric means Cmax of fluoxetine and norfluoxetine were determined when fluoxetine was administered alone (Day 24) and when fluoxetine was coadministered with LY2216684 (Day 27). The Day 27-to-Day 24 ratios of fluoxetine and norfluoxetine LS geometric means of Cmax and the associated 90% confidence interval (CI) of the ratios were calculated.
Time Frame: Predose and 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Days 24 and 27
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Arm/Group | LY2216684 + Fluoxetine
Number analyzed (Participants) | 20
nanogram per milliliter (ng/mL)
  fluoxetine alone | 160 [142 to 180]
  fluoxetine + LY2216684 | 160 [142 to 180]
  norfluoxetine alone | 144 [127 to 163]
  norfluoxetine + LY2216684 | 148 [131 to 168]
Statistical Analysis 1: Comparison: LY2216684 + Fluoxetine; Ratio of Geometric LS Means of Cmax for fluoxetine alone and fluoxetine + LY2216684; Test type: Superiority or Other; ANOVA; Ratio of Geometric LS Means = 1.00, 90% CI 2-sided [0.97 to 1.03]
Statistical Analysis 2: Comparison: LY2216684 + Fluoxetine; Ratio of Geometric LS Means of Cmax for norfluoxetine alone and norfluoxetine + LY2216684; Test type: Superiority or Other; ANOVA; Ratio of Geometric LS Means = 1.03, 90% CI 2-sided [1.00 to 1.07]

6. Secondary Outcome: Pharmacokinetic (PK) Parameter: Time to Maximum Plasma Concentration (Tmax) of Fluoxetine and Norfluoxetine
Description: Tmax of fluoxetine and norfluoxetine was determined using the median of paired differences between the 2 treatment groups when fluoxetine was administered alone (Day 24) and when fluoxetine was coadministered with LY2216684 (Day 27). The 90% confidence interval (CI) for the median of differences was calculated.
Time Frame: Predose and 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Days 24 and 27
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | LY2216684 + Fluoxetine
Number analyzed (Participants) | 20
hours
  fluoxetine alone | 6.00 [3.00 to 12.05]
  fluoxetine + LY2216684 | 6.00 [0.00 to 12.00]
  norfluoxetine alone | 12.00 [0.00 to 24.00]
  norfluoxetine + LY2216684 | 4.00 [0.00 to 12.00]
Statistical Analysis 1: Comparison: LY2216684 + Fluoxetine; Ratio of Geometric LS Means of Tmax for fluoxetine alone and fluoxetine + LY2216684; Test type: Superiority or Other; p = 0.4230, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.08, 90% CI 2-sided [-3.00 to 1.42]
Statistical Analysis 2: Comparison: LY2216684 + Fluoxetine; Ratio of Geometric LS Means of Tmax for norfluoxetine alone and norfluoxetine + LY2216684; Test type: Superiority or Other; p = 0.0293, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -4.00, 90% CI 2-sided [-6.50 to -1.00]

ADVERSE EVENTS:
Groups:
- LY2216684: LY2216684: 18 milligrams (mg) oral (po) once daily (QD) on Days 1-3 and Days 25-27.
Arm/Group | LY2216684 | Fluoxetine | LY2216684 + Fluoxetine
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 16/20 | 13/20 | 14/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2216684 (N=20) | Fluoxetine (N=20) | LY2216684 + Fluoxetine (N=20)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (8) | 4 (5) | 10 (10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (3) | 0 (0) | 5 (5)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 1 (1) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2) | 2 (4)
Headache (Nervous system disorders) | 1 (1) | 8 (12) | 4 (5)
Paraesthesia (Nervous system disorders) | 4 (4) | 0 (0) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Euphoric mood (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days